CLINICAL TRIAL: NCT03353701
Title: Effects of Experimentally-induced Reductions in Alcohol Consumption on Brain Cognitive and Clinical Outcomes, and Motivation for Changing Drinking in Older Persons With HIV Infection
Brief Title: 30-to-90 Day Challenge: Effects of Alcohol Cessation on Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other); Florida International University (Other); Brown University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CED000000011-N; U01AA020797-06 (NIH); U01AA026225 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-27 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Drinking; Chronic Inflammation; Neurocognitive Dysfunction; Liver Diseases; HIV Infections
MeSH Terms: conditions — Alcohol Drinking; Cognition Disorders; Liver Diseases; HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own controls with pre- and post-measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with or without HIV infection (Other): Participants will be asked to stop drinking for at least 30 and up to 90 days. The study will use Contingency Management (CM) with financial incentives to encourage participants to maximally reduce alcohol consumption.
  Interventions: Behavioral: Contingency Management (CM)

INTERVENTIONS:
Behavioral: Contingency Management (CM) — A reinforcement delivery method that involves financial incentive to participants for sustained alcohol abstinence. CM will start after the participants complete the baseline measures and last for at least 30 days and up to 90 days.

SUMMARY:
The objective for this project is to determine whether how certain behavioral and health functions change in persons with heavy drinking when they stop (or reduce) drinking for 30 days, and whether changes continue for up to 90 days. The study will also identify barriers and facilitators related to drinking reduction. The project will focus on clinical comorbidities including HIV disease control, cognitive and brain function, liver abnormalities, and chronic inflammation. The study teams propose to enroll 140 HIV+ and 40 HIV- adults with heavy drinking, and then use Contingency Management (CM) with financial incentives to encourage participants to maximally reduce alcohol consumption for 30 days. Participants will be required to wear an ankle biosensor (SCRAM monitor) at all times, which is used to monitor participants' drinking behavior. At 30 days, participants will complete a full day of follow-up, including cognitive testing, neuroimaging, blood testing, liver Fibroscan, and questionnaires. Many participants will also provide a stool sample for gut microbiome assessment at each time point. At 30 days, participants will participate in a motivational interview to discuss perceived benefits and obstacles to drinking reduction, and most participants will continue CM to 90 days (but can opt out at this point). Participants will complete another full-day assessment at 90 days, at which point persons may choose to drink or not on their own (no more CM). A final assessment will be conducted at 12 months. This A-B-A design will enable us to clearly identify whether alcohol effects on cognition and brain function are reversible in the context of HIV, and analyze specific cerebral and systemic pathophysiological factors contributing to these effects. The inclusion of HIV- adults will enable subgroup comparisons of alcohol reduction effects in the context of HIV vs. no-HIV. These HIV-negative participants will be recruited from the same settings as our HIV+ participants, and will include a similar proportion by age, race, and gender as the HIV+ participants. The study team will use information from the MI data and our other assessments to elucidate factors that predict both short term (during CM) and long-term (1-year) alcohol reductions, and study how changes in alcohol consumption affect important HIV clinical outcomes that will be monitored over time.

DETAILED DESCRIPTION:
This proposed study continues a line of research by Doctors Cohen, Cook, Kahler, and colleagues on heavy alcohol use, HIV-associated brain dysfunction, and long-term HIV outcomes. The study will build on our past findings to determine the extent to which marked reductions in alcohol consumption at 30 days and again at 90 days via contingency management (CM) improves cognitive-behavioral performance, underlying brain functions and pathophysiology, and HIV-associated health outcomes. This feature in itself is a novel contribution and has rarely been done, but more importantly, it reflects the mission of the collaboration to develop actionable data on clinical trajectories in HIV infected heavy drinkers over age 50 that will instill high confidence in guiding next therapeutic steps. The study team will obtain a better understanding of how persons with HIV stop drinking, and what factors influence long-term drinking changes. These important clinical and scientific questions need resolution for successful treatment and management of HIV+ adults. This study is motivated by evidence that HIV-associated neurocognitive dysfunction continues despite effective combined anti-retroviral therapies (cART). Even mild cognitive impairments have detrimental functional effects and health outcomes that worsen as HIV+ people age. Heavy alcohol consumption is common among HIV+ adults, and contributes to functional brain disturbances directly or indirectly via systemic metabolic or inflammatory disturbances. However, our past findings indicate that current alcohol use is more strongly associated with cognitive and brain dysfunction among HIV+ adults than lifetime consumption; and that adverse brain effects occur primarily with heavy drinking. Our overarching hypothesis is that the impact of ongoing heavy alcohol use on the brain and cognition may be reversible, providing a strong impetus for the proposed study. The study team will conduct our research in Florida, which has the highest number of new HIV infections in the US, as well as an increasingly diverse population with HIV+, 50% of whom are now aged 50 years or over in the state.

Our research will seek to modify alcohol consumption by using contingency management (CM) and measure for changes in brain pathophysiology and function, as well as changes in systemic inflammation, and gut and liver pathologies which are hypothesized pathways by which alcohol may increase brain dysfunction. The study team will also measure neurocognitive functioning related to learning, attention-executive functions, working memory, and processing speed, domains in which HIV+ persons experience persistent impairment. the study team will use Motivational Interviewing (MI) to learn more about how persons with and without HIV reduce drinking, what factors are associated with long-term drinking changes, and how these drinking changes influence HIV clinical health behavior and outcomes. If the impact of alcohol on systemic and cerebral inflammation is temporary, then reducing or eliminating alcohol consumption could dramatically improve cognitive function and indices of brain health, even among people who have consumed alcohol for many years in the past. Our research will directly test hypotheses that ongoing heavy alcohol consumption is associated with brain pathophysiology and inflammation that impairs both functioning and cognitive processing, and that the inflammation and its sequelae are reversible in most HIV+ persons with alcohol cessation. The proposed sample will be 140 adults with HIV infection and 40 adults without HIV infection (at least 25% female; age >50 years). Participants will be recruited from heavy drinkers (>=14 drinks/week women, >=21 drinks/week men) with HIV infection identified from our ongoing Florida Cohort. HIV- participants will be recruited from community medical clinics where flyers will be posted.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women;
2. Age: 50-75 yrs.;
3. 140 participants will have confirmed HIV (confirmed via baseline bloodwork) and 40 participants will be HIV negative
4. English speaking (will have protocol ready in Spanish in 2017);
5. Physically mobile;
6. Willing to participate in CM to reduce alcohol consumption, and to wear the alcohol biosensor for at least 30 days. All participants will be current, heavy drinkers (>=14 drinks/week women, >=21 drinks/week men), confirmed by baseline timeline follow-back, and by having evidence of at least 3 drinking episodes on the alcohol biosensor prior to baseline). Must blow a "zero" on breathalyzer at time of informed consent

Exclusion Criteria:

1. Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury).
2. Evidence of dementia (MOCA < 17).
3. Past opportunistic brain infection
4. Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis).
5. Current major psychiatric disturbance, including severe major depression.
6. Unstable medical conditions (e.g., cancer).
7. MRI contraindications (e.g., pregnancy, severe claustrophobia, metal implants).
8. Physical impairment precluding motor response or lying still.
9. Significant history of alcohol withdrawal as indicated by an Alcohol Withdrawal Symptom Checklist score ≥ 23 (within past year).
10. Unable to correctly answer a set of questions that demonstrate understanding of key aspects of the study, including the voluntary nature of the study, the purpose of the study, what participants are being asked to do as part of the study, and what are the risks related to participating in the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Neurocognitive Functions | Baseline, 30 Days
  Change in cognitive performance from baseline to 30-day follow-up. NIH Toolbox Cognition Battery is administered by a research assistant and consists of seven tests assessing memory, attention, cognitive flexibility, processing speed, and executive functioning. Summary scores will be calculated.

SECONDARY OUTCOMES:
Change in Neuroinflammation | Baseline, 30 Days
  Change in brain inflammation from baseline to 30-day follow-ups. Neuroinflammation is measured by cerebral metabolic neuroinflammatory markers, which include Magnetic Resonance Spectroscopy (MRS) metabolite concentrations (Cho and Myo-Inositol) and extracellular free water from Diffusor Tension Imaging sequences (DTI-FW).
Change in Brain Function | Baseline, 30 Days
  Change in Brain Function from baseline to 30-day follow-up. Brain function is measured by mean signal intensity for specific task-dependent brain regions from functional magnetic resonance imaging (fMRI).
Change in markers of systemic Inflammation | 30 Days
  Blood testing for biomarkers of systemic inflammation such as cytokines, ceramides, FIB-4, and marker of abnormal liver function.
Change in liver Status | 30 Days
  Evidence of liver fibrosis, fatty liver, and liver inflammation as measured by fibroscan
Change in Drinks/week in the Past 30 Days | Baseline, 1 Year
  Change in number of standard drinks per week in the past 30 days from baseline to 1 year follow-up, calculated from Timeline Follow Back (TLFB) interview.
Change in gut microbiome | Baseline, 30-days, 90-days, 1 year
  Change in the ratio of Firmicutes: Bacteriodetes ratio, and change in the relative abundance of Proteobacteria

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cook, Principal Investigator — University of Florida; Ronald Cohen, Principal Investigator — University of Florida
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited and de-identified datasets will be available to researchers after signing a data-use agreement with the University of Florida.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Our documents can be shared once the study begins. Data sharing will be an option for at least 5 years after the study is completed.
Access Criteria: Contact the principal investigator. In the future, information about how to request data will be on a public website
URL: http://sharc-research.org

REFERENCES:
- [Derived] Cook RL, Richards VL, Gullett JM, Lerner BDG, Zhou Z, Porges EC, Wang Y, Kahler CW, Barnett NP, Li Z, Pallikkuth S, Thomas E, Rodriguez A, Bryant KJ, Ghare S, Barve S, Govind V, Devieux JG, Cohen RA; 30-Day Challenge Research Team. Experimentally Induced Reductions in Alcohol Consumption and Brain, Cognitive, and Clinical Outcomes in Older Persons With and Those Without HIV Infection (30-Day Challenge Study): Protocol for a Nonrandomized Clinical Trial. JMIR Res Protoc. 2024 Apr 2;13:e53684. doi: 10.2196/53684. PMID 38564243
- [Derived] Richards VL, Wang Y, Porges EC, Gullett JM, Leeman RF, Zhou Z, Barnett NP, Cook RL. Using alcohol biosensors and biomarkers to measure changes in drinking: Associations between transdermal alcohol concentration, phosphatidylethanol, and self-report in a contingency management study of persons with and without HIV. Exp Clin Psychopharmacol. 2023 Dec;31(6):991-997. doi: 10.1037/pha0000637. Epub 2023 Jan 16. PMID 36649152